## **B-TREUH**

## NCT03787303

# Study of Euthyroid Hypothyroxinemia in Metastatic Breast Carcinoma Shruti Trehan, MD

April 14, 2022

### STATISTICAL ANALYSIS

#### **Statistical Methods**

- Compared mean scores over time to identify whether there were differences over time periods.
- ♦ Repeated measures analysis of variance (ANOVA) over 4 time periods to see if there was a statistical significance.